CLINICAL TRIAL: NCT01612195
Title: Success Rate, Continence, and Quality of Life With a Bioprosthetic Plug for Treating Complex Anal Fistula
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Unity Health Toronto (Other); Women's College Hospital (Other); St. Claraspital AG (Other); Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Michel Adamina, MD, PD, MSc, Senior Scientist, University Hospital, Basel, Switzerland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFP-2
Record Dates: First submitted 2012-06-02; First posted 2012-06-05 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Complex Anal Fistula
Keywords: anal fistula; anal continence; health-related quality of life
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anal fistula plug (Experimental)
  Interventions: Procedure: Anal fistula plug

INTERVENTIONS:
Procedure: Anal fistula plug — All patients have a draining seton for at least 6 weeks prior placement of the anal fistula plug. All patients are administered a general anesthetic and are operated in the lithotomy position. The seton is removed, but no curettage or irrigation of the fistula tract is performed. The plug is inserted through the internal opening, and pulled through the external opening until it fit snugly and its base is sutured to the internal sphincter with 2 interrupted 2-0 polyglactin 910 sutures. The tip of the plug is cut at skin level and not sutured. The external opening is left open to allow for drainage. The patient is instructed to restrict physical and sexual activity for 2 weeks postoperatively. Patients are seen in the post-operative clinic at 10 days, 6 weeks and 6 months as per protocol.
  Other Names: Anal fistula plug Surgisis®

SUMMARY:
Anal abscess-fistula disease is of common occurrence and has a significant impact on the quality of life of affected individuals. The course of abscess-fistula disease as well as its treatment modalities may affect anal continence. The present cohort study investigates the results of anal fistula plug surgery. In particular, this study focus on the impact of anal fistula plug surgery on fistula healing, quality of life, and anal continence. Fifty patients will be included and followed up at 6 weeks and 6 months after surgery in the clinic of participating surgeons.

DETAILED DESCRIPTION:
Anal abscess-fistula disease is of common occurrence and has a significant impact on the quality of life of affected individuals. The clinical course of abscess-fistula disease as well as its treatment modalities may affect anal continence. Anal fistula plug surgery is an Health Canada and FDA approved surgical treatment that has demonstrated promising results in terms of fistula healing and minimal patients' burden. The present cohort study prospectively investigates the results of anal fistula plug surgery performed in teaching hospitals affiliated to the University of Toronto. In particular, this study focus on the impact of anal fistula plug surgery on health-related quality of life, and its 2 major determinants anal continence and fistula healing. Fifty patients will be included and followed up at 6 weeks and 6 months after surgery in the clinic of participating surgeons. Quality of life and anal continence will be measured with the validated Short Form-36 Health Survey (SF-36 v2) and Fecal Incontinence Score Index (FISI) questionnaires, respectively. It is expected that the present study will provide objective information on the results and generalizability of anal fistula surgery, as well as on its impact on health-related quality of life and anal continence.

ELIGIBILITY:
Inclusion Criteria:

Complex anal fistula as defined by

* high transsphincteric fistula
* extrasphincteric fistula
* suprasphincteric fistula
* recurrent fistula
* multiple fistula openings, including horseshoe fistula
* imperfect continence- jeopardized anal continence (anterior transsphincteric fistula, prior anal surgery)

Exclusion Criteria:

* Uncomplicated fistula curable by simple fistulotomy
* History of inflammatory bowel disease
* Chronic immunosuppressive treatment (ie, systemic steroids for >3 days)
* Clinical heart failure as defined by a CCS angina severity class ≥ III
* Untreated cancer or cancer diagnosed/treated (all modalities) within 6 months
* Estimated life expectancy inferior to 6 months
* Incompetent subject
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Fistula healing | 6 months
  Clinical healing of a complex anal fistula as assessed in the clinic at 6 weeks and 6 months after anal fistula plug surgery. Further assessment prn.
Anal continence | 6 months
  Evaluation of anal continence by means of a validated questionnaire, namely the Fecal Incontinence Severity Index, at 6 weeks and 6 months after anal fistula plug surgery.
Quality of life | 6 months
  Evaluation of health-related quality of life by means of a validated questionnaire, namely the Short-Form 36 version 2, at 6 weeks and 6 months after anal fistula plug surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Adamina, MD, PD, MSc, Principal Investigator — University of Basel
Locations (1):
- University of Basel & Kantonsspital St.Gallen, Basel & St.Gallen, Switzerland